CLINICAL TRIAL: NCT04288414
Title: Prognostic Value for Predicting Outcome Using Functional Near-infrared Spectroscopy in Stroke Rehabilitation
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1601/332-003
Record Dates: First submitted 2019-07-16; First posted 2020-02-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- fNIRS applied: All of the participants' brain activity was evaluated with fNIRS.
  Interventions: Diagnostic Test: functional near-infrared spectroscopy

INTERVENTIONS:
Diagnostic Test: functional near-infrared spectroscopy — Functional near-infrared spectroscopy (fNIRS) is a non-invasive method that can evaluate the brain function by measuring the change in brain metabolic activity and hemodynamics during a given task with near-infrared spectroscopy.

SUMMARY:
To investigate the prognostic value of Functional Near-Infrared Spectroscopy (fNIRS) in stroke rehabilitation with serial measurements.

DETAILED DESCRIPTION:
Serial measurements (immediately after being transferred to rehabilitation department [T0], at discharge from inpatient rehabilitation [T1], and follow up at one to three months from stroke onset [T3]) using Functional Near-Infrared Spectroscopy (fNIRS) was done in all participants. The primary outcome was the outcome prediction rate using fNIRS parameter and clinical parameters. Secondary outcomes were as follows: fNIRS activation pattern, Laterality Index, Functional Connectivity, Fugl-Meyer Score, Modified Barthel Index, , Brunnstrom Stage, Box and Block Test, Grip Strength (handgrip, pinch grip, lateral prehension, three-jaw chuck), Modified Ashworth Scale (wrist flexor and extensor spasticity, elbow flexor, and extensor spasticity, long finger flexor spasticity), modified Rankin Scale score, Functional Ambulation Category, Glasgow Coma Scale, Neglect Evaluation Battery, Korean Version Western Aphasia Battery, and Scale for the Assessment and Rating of Ataxia.

The changes in the fNIRS measurements and clinical parameters will be analyzed and also the correlation between the two will be analyzed to identify the prognostic value of fNIRS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above.
* Diagnosed as stroke (infarction/hemorrhage) with imaging studies.
* Participants who have given consent after listening to the full explanations of this study.
* Able to understand the contents of this study and is able to sign to the written consent by his/herself.
* A legal representative has given written consent for those who meet the inclusion criteria but is unable to understand and agree by themselves due to impaired cognition, a legal representative.

Exclusion Criteria:

* Traumatic brain injury.
* Unable to perform simple commands (motor task during fNIRS scan) due to impaired cognition.
* Current symptoms are caused by diseases other than stroke (e.g., dementia, Parkinson's disease)
* Participants with any symptoms that may hinder the compliance or evaluation (e.g., delirium and agitation) process.
* Participants with any uncontrolled disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients who are receiving rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Outcome Prediction Rate | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Outcome prediction rate using fNIRS parameter and clinical parameters.

SECONDARY OUTCOMES:
Change of fNIRS activation pattern | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  The activation pattern was analyzed by nirsLAB software. This software provides data collection and correction function.
Change of Laterality Index | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  The formula for Laterality Index is (contralateral - ipsilateral)/(contralateral + ipsilateral). The range of Laterality index is -1 to 1. '-1' means all ipsilateral activation and '1' means all contralateral activation.
Change of National Institutes of Health Stroke Scale (NIHSS) Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Tool to quantify the impairment from stroke. On a scale from 0 to 42, 0 is one with no stroke symptoms and 42 is a stroke patient with the most severe symptoms. The 11 items of NIHSS are as follows: level of consciousness, horizontal eye movement, visual field test, facial palsy, motor arm, motor leg, limb ataxia, sensory, language, speech, and extinction and inattention.
Change of Glasgow Coma Scale (GCS) Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  A neurological scale to evaluate one's consciousness. There are three elements, which are eye response, verbal response, and motor response. A patient with best response will score 15 and a totally unresponsive patient will score 3.
Change of Modified Barthel Index (MBI) Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  The MBI is a scale that measures activities of daily living. It is composed of 10 categories: fecal incontinence, urinary incontinence, grooming, toilet use, feeding, transfers (e.g., from chair to bed), walking, dressing, climbing stairs, and bathing. A higher score is a patient with better ability to live independently.
Fugl-Meyer Assessment (FMA) Scale | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  A scale that assess the impairment in a stroke patient. It has three points for each item. When a patient can perform a given task fully, 2 point is given. 1 point is given for partial performance and 0 for not being able to perform the task. The five domains of FMA scale are: motor function (Maximum score in upper limb = 66, Maximum score in lower limb = 34), sensory function (Maximum score = 24), balance (Maximum score = 14), range of motion of joints (Maximum score = 44), and joint pain (Maximum score = 44).
Change of Brunnstrom Stage Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Staging of recovery from stroke. The stages are: 1. flaccidity, 2. developing spasticity, 3. pronounced spasticity, 4. spasticity and influence of synergies start to decrease, 5. spasticity declines even more, and 6. no spasticity and near normal stage.
Change of Box and Block Test Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  A test using a box and and blocks to evaluate the upper extremity function.
Change of Grip strength | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Used JAMAR Hydraulic Hand Dynamometer and JAMAR Hydraulic Pinch Gauge. Hand grip, pinch grip, lateral prehension, and three jaw chuck were measured.
Change of Modified Ashworth Scale Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Measurement of spasticity during passive stretching. Wrist flexor/extensor spasticity, elbow flexor/extensor spasticity, and long finger flexor spasticity were measured. On a scale of 0 to 4, 0 means there is no spasticity and 4 means it is rigid in flexion or extension.
Change of Modified Rankin Scale (mRS) Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  A popular validated functional outcome measure in stroke. On a scale from 0 to 6, 0 is one with no symptom and 6 is the worst meaning death.
Change of Functional Ambulatory Category (FAC) Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  On a scale from 1 to 6 ambulation status is described. 1 being the worst and 6 being independent at level and non-level surfaces also.
Change of Neglect Evaluation Battery Score | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Includes Motor Free Visual Perception Test (MVPT), Line Bisection Test, Albert Test, Clock Drawing, Comb and Razor, and Catherine Bergego Scale. Used electrical method if available. Otherwise test was performed.
Change of Western Aphasia Battery (WAB) | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Measures aphasia type and severity
Change of Scale for the Assessment and Rating of Ataxia (SARA) | After 2-3 weeks from stroke onset (T0), Immediately after 2-3 weeks of rehabilitation (T1), After 1-3 months from stroke onset (T2)
  Clinical scale that assess different impairments in cerebellar ataxia. Consisted of 8 items. It is related to gait, stance, sitting, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, Ph.D, Principal Investigator — Seoul National University Bundang Hospital, Seongnam, South Korea
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No